CLINICAL TRIAL: NCT01423110
Title: A Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of BYM338 in Patients With Sporadic Inclusion Body Myositis
Brief Title: Efficacy, Safety and Tolerability of BYM338 in Patients With Sporadic Inclusion Body Myositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338X2205
Record Dates: First submitted 2011-08-12; First posted 2011-08-25 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-02

CONDITIONS: Sporadic Inclusion Body Myositis
Keywords: sporadic Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BYM338 (Experimental)
  Interventions: Biological: BYM338
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BYM338
  Arms: BYM338
Biological: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety and tolerability of BYM338 in patients with sporadic Inclusion Body Myositis

ELIGIBILITY:
Inclusion Criteria:

- Males and Females aged 40-80 with a confirmed diagnosis of sporadic Inclusion Body Myositis

Exclusion Criteria:

* Unable to walk at least 3 meters without assistance from another person
* Use of oral beta agonists, oral corticosteroids, androgens or androgen inhibitors, or intravenous gamma globulin in the last 6 months
* patients with a history or presence of renal impairment and/or liver disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of BYM338 on Thigh Muscle Volume by MRI | 8 weeks
  Change in thigh muscle volume

SECONDARY OUTCOMES:
Effect of BYM338 on muscle function by 'Timed Get Up and Go' test | 8 weeks
  Change in muscle function measured on scale by test results

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Boston, Massachusetts

REFERENCES:
- [Result] Amato AA, Sivakumar K, Goyal N, David WS, Salajegheh M, Praestgaard J, Lach-Trifilieff E, Trendelenburg AU, Laurent D, Glass DJ, Roubenoff R, Tseng BS, Greenberg SA. Treatment of sporadic inclusion body myositis with bimagrumab. Neurology. 2014 Dec 9;83(24):2239-46. doi: 10.1212/WNL.0000000000001070. Epub 2014 Nov 7. PMID 25381300
- See also: Results for CBYM338X2205 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10243